CLINICAL TRIAL: NCT05104268
Title: A Randomized Study of a New Medical Device for Oral Mucositis (MDOM Trial)
Brief Title: Study of a New Medical Device for Oral Mucositis
Acronym: MDOM
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Unable to recruit due to the relatively infrequent occurrence of oral mucositis
Sponsor: E2Bio Life Sciences, LLC (Industry)
Collaborators: Hematology Center after Prof. R. Yeolyan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BL001
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Oral Mucositis; Stem Cell Transplant Complications
Keywords: Stem Cell Transplantation; Oral Mucositis; Cancer; Complications of chemotherapy; Oral Inflammation; Oral Pain; Pharmacokinetics; Oral Topical Therapy; Oral Inserted Device; Oral Resonance Time
MeSH Terms: conditions — Stomatitis; Neoplasms

STUDY DESIGN:
Intervention Model Description: Subjects will then be randomized into two groups. Group 1 will continue standard therapy with oral topical agents for oral mucositis. Group 2 will additionally receive Bocaliner™ devices along with cleaning materials with instructions about device use and cleaning. Subjects in the Group 2 will use Bocaliner™ with each topical treatment for oral mucositis up to 5 times per day for 2 weeks or shorter if not tolerated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard Therapy (Active Comparator): Subjects will then be randomized into two groups. The Standard Therapy Group will continue their usual therapy with oral topical agents for oral mucositis.
  Interventions: Device: Bocaliner
- Bocaliner (Experimental): Participants that are randomized to the Bocaliner Group will place Bocaliner™ inside of their mouth for 5 minutes and fill out the Initial Bocaliner™ Questionnaire. They will then continue all original therapy for oral mucositis, including oral topical treatments and general hygiene, and will place the Bocaliner™ device inside of their mouth and hold it in place up to 40 minutes as instructed after each topical treatment.
  Interventions: Device: Bocaliner

INTERVENTIONS:
Device: Bocaliner — Bocaliner is an orally inserted device that is held within the mouth following the administration of mouthwashes, gels, and rinses that are used to treat pain associated with oral mucositis, and to reduce inflammation and to accelerate healing of oral mucositis.
  Other Names: Standard Treatments for Oral Mucositis

SUMMARY:
This is a single-center randomized controlled trial of a new medical device (Bocaliner™) that has been designed to improve the treatment of chemotherapy-induced oral mucositis in patients undergoing cancer treatment. The goal of this study is to determine tolerance and response to the use of Bocaliner™ as reported by patients with chemotherapy and/or radiation therapy-induced oral mucositis.

DETAILED DESCRIPTION:
All patients will be referred by their treating physicians to the designated study healthcare providers. Patients will have been diagnosed with oral mucositis and will be receiving oral topical medication for oral pain as well as other problems related to oral mucositis. All subjects will sign an informed consent form.

Initially, subjects will undergo an oral examination and for determination of the World Health Organization (WHO) Oral Toxicity Scale and will then complete a General Oral Mucositis Assessment Scale.

Subjects will then be randomized into two groups. Group 1 will continue standard therapy with oral topical agents for oral mucositis. Group 2 will additionally receive Bocaliner™ devices along with cleaning materials with instructions about device use and cleaning. Subjects in the Group 2 will use Bocaliner™ with each topical treatment for oral mucositis up to 5 times per day for 2 weeks or shorter if not tolerated.

Subjects assigned to the Group 1 will continue the original therapy for oral mucositis, including oral topical treatments and general hygiene measures. Participants that are randomized to the Group 2 will place Bocaliner™ inside of their mouth for 5 minutes and fill out the Initial Bocaliner™ Questionnaire. They will then continue all original therapy for oral mucositis, including oral topical treatments and general hygiene, and will place the Bocaliner™ device inside of their mouth and hold it in place up to 40 minutes as instructed after each topical treatment.

All subjects will be contacted by the Research Coordinator via phone call at 5 and 10 days after the initial enrollment and invited to answer the questions from the Modified PROMS Questionnaire at the hospital. Alternatively, the questionnaire can be provided via email, or the questions can be answered via phone call, if preferred by a patient. Subjects in Group 2 will describe their experience of using Bocaliner™ through the Bocaliner™ Follow-up Questionnaire. All subjects will give a detailed description of their current medication usage for oral mucositis. Participants from both groups will return to their practitioners after 14 days and undergo a general oral examination. The WHO Oral Toxicity Scale will be used to assess the grade of oral mucositis. Subjects will also complete the Modified PROMS Questionnaire at days 5, 10, and 14 to understand the impact of standard treatment vs Bocaliner™ on symptoms related to oral mucositis.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic chemotherapy-induced oral mucositis
* Need for oral topical therapy for symptomatic treatment
* Absence of other chronic oral disorders
* Properly obtained written informed consent
* Age of 18 years or older
* Patient is willing to use the Bocaliner™ device for 2 weeks
* No concurrent use of medications modulating pain

Exclusion Criteria:

* Chronic oral conditions other than chemotherapy-induced oral mucositis
* No informed consent
* Age of <18
* Inability to place the device in his/her mouth and keep it in place for at least 10 minutes due to severe oral pain, large lesions, or any other reason
* Inability/unwillingness to wear Bocaliner™ for the study period
* Concurrent use of pain-modulating agents
* Individuals with known allergies to silicone materials
* Individuals with severe difficulties to communicate and understand

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Patient-Reported Oral Mucositis Symptom (The Modified PROMS Questionnaire) Pain Score | 5, 10, and 14 days
  The modified PROMS score is designed to measure symptoms and quality of life in patients with oral mucositis. It consists of twelve questions. The range in scores for each section is 0 to 100. Higher scores on the Modified PROMS indicate worse outcomes.
  The range in the Pain Score of the Modified PROMS Questionnaire is from 0 to 100.

SECONDARY OUTCOMES:
Change in other symptoms of oral mucositis on the Patient-Reported Oral Mucositis Symptom (The Modified PROMS Questionnaire. | 5, 10, and 14 days
  The modified PROMS score is designed to measure symptoms and quality of life in patients with oral mucositis. It consists of twelve questions. The range in scores for each question is 0 to 100. Higher scores on the PROMS Questionnaire indicate worse outcomes.
Change of oral mucositis grade in the World Health Organization Grade,(WHO Mucositis Grade) | 5, 10, and 14 days
  The WHO Mucositis grade is based on the appearance of the oral mucosa and the effect of oral mucositis on nutritional intake. The range of grades is from 1 to 4. Higher WHO Mucositis grades indicate worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Yervand Hakoban, MD PhD, Principal Investigator — Hematology Center after Prof. R. Yeolyan, MH RA
Locations (1):
- Hematology Center after Prof. R. Yeolyan MH RA, Yerevan, Armenia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be available to other research scientists who meet screening criteria by principal investigator.
Supporting Information: CSR
Time Frame: January 2023 through January 2024
Access Criteria: 1. Data scientists from accredited clinical organizations
  2. Accepted review by principal investigator for the planned purpose for data use

REFERENCES:
- [Result] Jones JA, Avritscher EB, Cooksley CD, Michelet M, Bekele BN, Elting LS. Epidemiology of treatment-associated mucosal injury after treatment with newer regimens for lymphoma, breast, lung, or colorectal cancer. Support Care Cancer. 2006 Jun;14(6):505-15. doi: 10.1007/s00520-006-0055-4. Epub 2006 Apr 7. PMID 16601950
- [Result] Lalla RV, Bowen J, Barasch A, Elting L, Epstein J, Keefe DM, McGuire DB, Migliorati C, Nicolatou-Galitis O, Peterson DE, Raber-Durlacher JE, Sonis ST, Elad S; Mucositis Guidelines Leadership Group of the Multinational Association of Supportive Care in Cancer and International Society of Oral Oncology (MASCC/ISOO). MASCC/ISOO clinical practice guidelines for the management of mucositis secondary to cancer therapy. Cancer. 2014 May 15;120(10):1453-61. doi: 10.1002/cncr.28592. Epub 2014 Feb 25. PMID 24615748
- [Result] Chaudhry HM, Bruce AJ, Wolf RC, Litzow MR, Hogan WJ, Patnaik MS, Kremers WK, Phillips GL, Hashmi SK. The Incidence and Severity of Oral Mucositis among Allogeneic Hematopoietic Stem Cell Transplantation Patients: A Systematic Review. Biol Blood Marrow Transplant. 2016 Apr;22(4):605-616. doi: 10.1016/j.bbmt.2015.09.014. Epub 2015 Sep 26. PMID 26409924
- [Result] Sio TT, Le-Rademacher JG, Leenstra JL, Loprinzi CL, Rine G, Curtis A, Singh AK, Martenson JA Jr, Novotny PJ, Tan AD, Qin R, Ko SJ, Reiter PL, Miller RC. Effect of Doxepin Mouthwash or Diphenhydramine-Lidocaine-Antacid Mouthwash vs Placebo on Radiotherapy-Related Oral Mucositis Pain: The Alliance A221304 Randomized Clinical Trial. JAMA. 2019 Apr 16;321(15):1481-1490. doi: 10.1001/jama.2019.3504. PMID 30990550
- [Result] Kushner JA, Lawrence HP, Shoval I, Kiss TL, Devins GM, Lee L, Tenenbaum HC. Development and validation of a Patient-Reported Oral Mucositis Symptom (PROMS) scale. J Can Dent Assoc. 2008 Feb;74(1):59. PMID 18298885